CLINICAL TRIAL: NCT02046837
Title: A Pilot RCT and Economic Analysis of Three Exercise Delivery Methods in Men With Prostate Cancer on ADT
Brief Title: An Exercise Trial and Economic Analysis in Men With Prostate Cancer
Acronym: ADT Ex RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UHN ADT Ex 01
Record Dates: First submitted 2014-01-20; First posted 2014-01-28 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Exercise; Elderly; Quality of life; Fatigue; Physical fitness; Adherence; Cost-effectiveness
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Supervised 1:1 exercise (Experimental): This intervention arm will include 3 one-on-one, supervised sessions per week for 6 months with a certified exercise specialist. Flexibility training will include stretching for 5-10 minutes at the beginning and end of each session. Aerobic training will involve 30 minutes of low-impact step aerobics. Resistance training will be conducted using resistance bands, a stability ball, and an exercise mat with 8 prescribed exercises that target the major muscle groups. Participants will be encouraged to perform exercises independently on additional days, for a total of 4-5 days per week of exercise.
  Interventions: Behavioral: Supervised 1:1 exercise
- Supervised group exercise (Experimental): This intervention arm will include 3 group, supervised sessions per week for 6 months with a certified exercise specialist. Supervised sessions will be delivered in a group format with 4-8 participants per group. Flexibility training will include stretching for 5-10 minutes at the beginning and end of each session. Aerobic training will involve 30 minutes of low-impact step aerobics. Resistance training will be conducted using resistance bands, a stability ball, and an exercise mat with 8 prescribed exercises that target the major muscle groups. Participants will be encouraged to perform exercises independently on additional days, for a total of 4-5 days per week of exercise.
  Interventions: Behavioral: Supervised group exercise
- Home-based exercise (Experimental): The same protocol and training frequency as the supervised programs described above will be followed. However, all exercises will be completed independently by participants. Specific exercises in the aerobic program may be modified to accommodate patient preference (same target heart rate range as supervised groups). Participants will be supported with smartphone technology and remote 'health coaches' during the intervention phase. This will help to ensure participant adherence, appropriate progression, and safety.
  Interventions: Behavioral: Home-based exercise

INTERVENTIONS:
Behavioral: Supervised 1:1 exercise — The exercise program will be delivered in a personal training (1:1) format by a certified exercise specialist.
  Arms: Supervised 1:1 exercise
Behavioral: Supervised group exercise — The exercise program will be delivered in a group format (4-8 participants per group) by a certified exercise specialist.
  Arms: Supervised group exercise
Behavioral: Home-based exercise — The exercise program will be executed independently by participants in a home-based setting. Home-based participants will be supported with remote health coaching and smartphone technology.
  Arms: Home-based exercise

SUMMARY:
Prostate Cancer (PC) affects 1 in 7 men. Nearly half of those diagnosed with PC will receive androgen deprivation therapy (ADT) as part of their treatment. ADT is good at managing PC but has many side effects. Researchers have shown that exercise, specifically one-on-one supervised exercise improves many of the side effects of ADT. However, exercise programs for men on ADT are not widely available. More questions need to be answered in order for exercise programs to become part of PC treatment. First, can programs that require fewer resources, such as group-exercise or home-based exercise, also improve ADT side-effects? Second, do exercise-related benefits continue beyond the structured exercise program? And what makes people continue exercising? Third, which exercise program is most cost-effective?

In this study, the investigators will compare: (a) group supervised in-centre; (b) home-based supported; and (c) 1:1 supervised in-centre exercise programs to see which program is most effective for men with PC on ADT. The investigators will also look at what motivates people to continue to exercise both during a structured program and after the program is complete and will examine which exercise program is most cost-effective.

The investigators will ask men with PC on ADT that are being treated at either Princess Margaret Cancer Centre in Toronto or the Tom Baker Cancer Centre in Calgary to participate in the study. When a patient agrees to participate, he will be randomly placed in 1 of the 3 exercise programs. All programs will include the same type of exercises (aerobic, resistance and flexibility) and all participants will exercise 4-5 days per week for 30 minutes per day (as tolerated) for the length of the program (6 months). The investigators will look at how men with PC on ADT respond to the exercise program by measuring quality of life (QOL), fatigue and different physical measures before, during, and after the exercise program.

Although the investigators know that supervised one-on-one exercise is most effective at improving ADT side-effects, it is unknown if other forms of exercise are just as beneficial and more financially responsible. This study will allow the investigators to begin to answer these questions so that structured exercise programs become a regular part of PC treatment.

ELIGIBILITY:
Inclusion Criteria:

* confirmed prostate cancer
* starting or continuing on ADT for at least 6 months
* fluent in English
* able to provide consent
* live close to a study centre
* screened with the Physical Activity Readiness Questionnaire (PAR-Q+ or PARmed-X) to ensure safe exercise participation OR receive medical clearance by attending physician

Exclusion Criteria:

* already meeting guidelines for moderate to vigorous physical activity (MVPA) as defined by the Canadian Physical Activity Guidelines (greater than or equal to 150 minutes of MVPA per week)
* conditions that would interfere with ability to participate

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in health-related quality of life (QOL) at 3, 6, 9, and 12 months | Every 3 months for 1 year
  Measured by the Functional Assessment of Cancer Therapy-General (FACT-G), health-related QOL refers to those aspects of QOL that relate a person's health to their physical, functional, psychological, and social well-being. The FACT-G is a well-validated and widely used QOL measure. It can be completed in 8-10 minutes and has published normative data.

SECONDARY OUTCOMES:
Change from baseline in quality of life (QOL) at 3, 6, 9, and 12 months | Every 3 months for 1 year
  Supplementing the assessment of health-related QOL, prostate-specific QOL will be measured with the FACT-P. The FACT-P contains 12 prostate-specific items covering domains of urinary function, sexual function, pain, and related symptoms. It is well-validated and used in multiple prior exercise trials.
Change from baseline in fatigue at 3, 6, 9, and 12 months | Every 3 months for 1 year
  The FACT-Fatigue (FACT-F), includes 13 items measuring cancer-related fatigue. It has excellent reliability and validity. Fatigue is a common symptom in men on ADT and has been shown to benefit from exercise.
Change from baseline in aerobic fitness (VO2peak) at 3, 6, 9, and 12 months | Every 3 months for 1 year
  Aerobic fitness will be assessed using a treadmill-based graded exercise test (modified Bruce protocol) to maximal exertion. Standard test termination criteria apply.
Change from baseline in musculoskeletal fitness at 3, 6, 9, and 12 months | Every 3 months for 1 year
  Musculoskeletal fitness will be assessed using a sit-to-stand test, a common, simple, and validated measure of functional lower body strength.
Change from baseline in grip strength at 3, 6, 9, and 12 months | Every 3 months for 1 year
  Grip strength is a measure of upper body strength and is responsive to ADT use. It predicts long-term disability and mortality in middle-aged and older adults.
Change from baseline in body composition at 6 and 12 months | Every 6 months for 1 year
  Body composition will be assessed via bioelectrical impedance analysis (BIA), waist circumference (WC), WC:hip ratio, and BMI, following the standardized Canadian Society for Exercise Physiology protocol.
Change from baseline in bone mineral density at 12 months | Baseline and 1 year.
  Bone mineral density (lumbar spine, hip, femoral neck, and distal 1/3 radius) will be assessed using dual x-ray absorptiometry (DXA).
Change from baseline in biological outcomes at 6 and 12 months | Every 6 months for 1 year
  Insulin sensitivity and blood lipid profiles have been shown to be negatively affected by ADT. To examine the effect of exercise on these metabolic outcomes, fasting lipids and blood glucose, in addition to PSA level, will be assessed. Serum banking will also be done for use in future studies.
Change from baseline in adherence predictors at 3, 6, 9, and 12 months | Every 3 months for 1 year
  We will use a social ecological approach to assess factors at three related levels using the following validated measures: Exosystem Measures: Neighborhood Environment Walkability Scale: Short Form (NEWS-A); Mesosystem Measures: Health Care Climate Questionnaire (HCCQ short form) and Relatedness to Others in Physical Activity scale; Microsystem Measures: Behavioral Regulations in Exercise Questionnaire-2 (BREQ-2) and a Planning, Attitudes, & Barriers scale. Time spent in activities that are characterized by an energy expenditure ≤ 1.5 metabolic equivalents and a sitting or reclining posture will be assessed using the Sedentary Behaviour Questionnaire that is used in large cohort studies and has demonstrated evidence of reliability and validity.
Change from baseline in cost-effectiveness at 3, 6, 9, and 12 months | Every 3 months for 1 year
  We will collect economically relevant data about health status using preference-based (utility) instruments (EQ-5D). Productivity losses and out-of-pocket expenditures, in addition to hospitalization, drug co-pay, and health visit data will be gathered using a patient questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir MH Alibhai, MD, MSc, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - University of Calgary/Tom Baker Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Papadopoulos E, Leach HJ, Tomlinson G, Durbano S, Danyluk JM, Sabiston CM, Mina DS, Alibhai SMH, Culos-Reed SN. Factors predicting gains in moderate-to-vigorous physical activity in prostate cancer survivors on androgen deprivation therapy. Support Care Cancer. 2022 Nov;30(11):9011-9018. doi: 10.1007/s00520-022-07300-2. Epub 2022 Aug 10. PMID 35948848
- [Derived] Alibhai SMH, Santa Mina D, Ritvo P, Tomlinson G, Sabiston C, Krahn M, Durbano S, Matthew A, Warde P, O'Neill M, Timilshina N, Segal R, Culos-Reed N. A phase II randomized controlled trial of three exercise delivery methods in men with prostate cancer on androgen deprivation therapy. BMC Cancer. 2019 Jan 3;19(1):2. doi: 10.1186/s12885-018-5189-5. PMID 30606137
- [Derived] Alibhai SM, Santa Mina D, Ritvo P, Sabiston C, Krahn M, Tomlinson G, Matthew A, Segal R, Warde P, Durbano S, O'Neill M, Culos-Reed N. A phase II RCT and economic analysis of three exercise delivery methods in men with prostate cancer on androgen deprivation therapy. BMC Cancer. 2015 Apr 25;15:312. doi: 10.1186/s12885-015-1316-8. PMID 25908311